CLINICAL TRIAL: NCT03801525
Title: Phase 2/3 Randomized Study to Assess the Efficacy and Safety of Ublituximab in Combination With Umbralisib and Venetoclax (U2-V) Compared to Ublituximab and Umbralisib (U2) in Subjects With Chronic Lymphocytic Leukemia (CLL)
Brief Title: Study to Assess the Efficacy and Safety of Ublituximab in Combination With Umbralisib and Venetoclax Compared to Ublituximab in Combination With Umbralisib in Subjects With CLL (ULTRA-V)
Acronym: ULTRA-V
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Strategic/Business decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U2-VEN-207
Record Dates: First submitted 2019-01-09; First posted 2019-01-11 (Actual); Results first posted 2024-04-19 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: CLL; SLL
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ublituximab; umbralisib; venetoclax

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) (Experimental): Participants were administered ublituximab, 150 milligrams (mg), intravenous (IV) infusion on Day 1, 750 mg on Day 2, 900 mg on Days 8 and 15 of Cycle 1, followed by 900 mg on Day 1 of Cycles 2-6; umbralisib, 800 mg, oral tablet, once daily (QD) through Cycles 1-24; venetoclax, oral tablet, QD, 20 mg on Days 1-7, 50 mg on Days 8-14, 100 mg on Days 15-21, 200 mg on Days 22-28 of Cycle 4, followed by 400 mg on Days 1-28 of Cycles 5-24. MRD positive participants were administered umbralisib, 800 mg, oral tablet, QD, on Days 1-28 from Cycle 25 onwards (1 Cycle = 28 days), until disease progression, unacceptable toxicity, or withdrawal from the study.
  Interventions: Drug: Ublituximab; Drug: Umbralisib; Drug: Venetoclax
- Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) (Experimental): Participants were administered ublituximab, 150 mg, IV infusion on Day 1, 750 mg on Day 2, 900 mg on Days 8 and 15 of Cycle 1, followed by 900 mg on Day 1 of Cycles 2-6, 9,12, and 15; umbralisib, 800 mg, oral tablet, QD through Cycles 1-15; venetoclax, oral tablet, QD, 20 mg on Days 1-7, 50 mg on Days 8-14, 100 mg on Days 15-21, 200 mg on Days 22-28 of Cycle 4, followed by 400 mg on Days 1-28 of Cycles 5-15 (1 Cycle = 28 days).
  Interventions: Drug: Ublituximab; Drug: Umbralisib; Drug: Venetoclax
- Phase 3: Ublituximab + Umbralisib (U2) (Experimental): Participants were administered ublituximab, 150 mg, IV infusion on Day 1, 750 mg on Day 2, 900 mg on Days 8 and 15 of Cycle 1, followed by 900 mg on Day 1 of Cycles 2-6, then every three cycles along with umbralisib, 800 mg, oral tablet, QD (1 Cycle = 28 days) from Cycle 1 until disease progression, unacceptable toxicity, or withdrawal from the study.
  Interventions: Drug: Ublituximab; Drug: Umbralisib

INTERVENTIONS:
Drug: Ublituximab — * recombinant chimeric anti-CD20 (cluster of differentiation 20) monoclonal antibody
  * administered as an IV infusion
  Other Names: TG-1101
Drug: Umbralisib — * inhibitor of phosphoinositide 3-kinase (PI3K) delta and casein kinase 1 epsilon (CK1e)
  * Tablet form
  Other Names: TGR-1202; UKONIQ
Drug: Venetoclax — * B-cell lymphoma 2 (BCL-2) inhibitor
  * Tablet form
  Other Names: Venclexta®
  Arms: Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V); Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V)

SUMMARY:
ULTRA-V: Study to Assess the Efficacy and Safety of Ublituximab in Combination with Umbralisib and Venetoclax (U2-V) Compared to Ublituximab and Umbralisib (U2) in Subjects with Chronic Lymphocytic Leukemia (CLL)

DETAILED DESCRIPTION:
This is an open-label, multicenter, Phase 2/3 study to evaluate the efficacy and safety of the combination of ublituximab + umbralisib + venetoclax (U2-V) compared to the combination of ublituximab + umbralisib (U2) in participants with either treatment naïve or previously treated CLL/ small lymphocytic lymphoma (SLL).

ELIGIBILITY:
Inclusion Criteria:

* Chronic lymphocytic leukemia (CLL)/ small lymphocytic lymphoma (SLL) that warrants treatment
* Adequate organ system function as specified in the protocol
* Ability to follow protocol procedures.

Exclusion Criteria:

* Subjects receiving cancer therapy or any investigational drug within 21 days of Cycle 1, Day 1
* Prior exposure to any PI3K inhibitor or venetoclax
* Autologous hematologic stem cell transplant within 6 months of study entry. Prior allogeneic hematologic stem cell transplant is excluded
* Active Hepatitis B or Hepatitis C.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 277 (Actual)
Dates: Start 2019-05-16 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (48):
- United States (48):
  - TG Therapeutics Investigational Trial Site, Birmingham, Alabama
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Tucson, Arizona
  - TG Therapeutics Investigational Trial Site, Duarte, California
  - TG Therapeutics Investigational Trial Site, La Jolla, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Stamford, Connecticut
  - TG Therapeutics Investigational Trial Site, Boca Raton, Florida
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, Jacksonville, Florida
  - TG Therapeutics Investigational Trial Site, St. Petersburg, Florida
  - TG Therapeutics Investigational Trial Site, Tampa, Florida
  - TG Therapeutics Investigational Trial Site, Atlanta, Georgia
  - TG Therapeutics Investigational Trial Site, Decatur, Illinois
  - TG Therapeutics Investigational Trial Site, Niles, Illinois
  - TG Therapeutics Investigational Site, Peoria, Illinois
  - TG Therapeutics Investigational Trial Site, Fort Wayne, Indiana
  - TG Therapeutics Investigational Trial Site, Indianapolis, Indiana
  - TG Therapeutics Investigational Trial Site, Des Moines, Iowa
  - TG Therapeutics Investigational Trial Site, Westwood, Kansas
  - TG Therapeutics Investigational Site, Louisville, Kentucky
  - TG Therapeutics Investigational Trial Site, Bethesda, Maryland
  - TG Therapeutics Investigational Trial Site, Columbia, Maryland
  - TG Therapeutics Investigational Trial Site, Ann Arbor, Michigan
  - TG Therapeutics Investigational Trial Site, Detroit, Michigan
  - TG Therapeutics Investigational Trial Site, Rochester, Minnesota
  - TG Therapeutics Investigational Trial Site, Omaha, Nebraska
  - TG Therapeutics Investigational Trial Site, Lebanon, New Hampshire
  - TG Therapeutics Investigational Trial Site, Hackensack, New Jersey
  - TG Therapeutics Investigational Trial Site, Morristown, New Jersey
  - TG Therapeutics Investigational Trial Site, New York, New York
  - TG Therapeutics Investigational Trial Site, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, Columbus, Ohio
  - TG Therapeutics Investigational Trial Site, Eugene, Oregon
  - TG Therapeutics Investigational Trial Site, Philadelphia, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Charleston, South Carolina
  - TG Therapeutics Investigational Trial Site, Greenville, South Carolina
  - TG Therapeutics Investigational Trial Site, Chattanooga, Tennessee
  - TG Therapeutics Investigational Trial Site, Knoxville, Tennessee
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Austin, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Tyler, Texas
  - TG Therapeutics Investigational Trial Site, Ogden, Utah
  - TG Therapeutics Investigational Trial Site, Salt Lake City, Utah
  - TG Therapeutics Investigational Trial Site, Blacksburg, Virginia
  - TG Therapeutics Investigational Trial Site, Gainesville, Virginia
  - TG Therapeutics Investigational Trial Site, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 277 participants were enrolled at investigative sites in the United States from 16 May 2019 to 20 December 2022.
Period: Overall Study
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
Started | 165 | 56 | 56
Intent-To-Treat (ITT) Population (In Phase 2, ITT population consisted of all participants who received at least one dose of each study drug (ublituximab, umbralisib, and venetoclax); and in Phase 3, ITT population consisted of all participants who were randomized.) | 149 | 56 | 56
Completed | 11 | 0 | 0
Not Completed | 154 | 56 | 56
Not completed — Adverse Event | 17 | 1 | 0
Not completed — Conditions Requiring Therapeutic Intervention Not Permitted by The Protocol | 1 | 0 | 0
Not completed — Death | 29 | 1 | 4
Not completed — Disease Progression | 6 | 0 | 1
Not completed — Inability to Comply With Study Requirements | 1 | 1 | 0
Not completed — Investigator Decision | 18 | 1 | 0
Not completed — Minimal Residual Disease (MRD) Negativity and Tumor Response | 14 | 0 | 0
Not completed — Sponsor Discontinuation of the Study | 24 | 49 | 43
Not completed — Started Non-protocol Anti-cancer Therapy | 2 | 1 | 3
Not completed — Withdrawal of Subject Consent | 38 | 2 | 1
Not completed — Reason not Specified | 4 | 0 | 4

BASELINE CHARACTERISTICS:
Population: Safety population consisted of all participants who received at least one dose of any study drug (ublituximab, umbralisib, and venetoclax).
Groups:
- Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V): Participants were administered ublituximab, 150 mg, IV infusion on Day 1, 750 mg on Day 2, 900 mg on Days 8 and 15 of Cycle 1, followed by 900 mg on Day 1 of Cycles 2-6; umbralisib, 800 mg, oral tablet, QD through Cycles 1-24; venetoclax, oral tablet, QD, 20 mg on Days 1-7, 50 mg on Days 8-14, 100 mg on Days 15-21, 200 mg on Days 22-28 of Cycle 4, followed by 400 mg on Days 1-28 of Cycles 5-24. MRD positive participants were administered umbralisib, 800 mg, oral tablet, QD, on Days 1-28 from Cycle 25 onwards (1 Cycle = 28 days), until disease progression, unacceptable toxicity, or withdrawal from the study.
- Total: Total of all reporting groups
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2) | Total
Number analyzed (Participants) | 165 | 56 | 53 | 274
Age, Continuous [Mean (Full Range); unit: years] | 65.9 [44 to 85] | 65.5 [46 to 91] | 62.9 [38 to 80] | 65.3 [38 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 60 | 22 | 14 | 96
  Male | 105 | 34 | 39 | 178
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 2 | 1 | 8
  Not Hispanic or Latino | 158 | 53 | 49 | 260
  Unknown or Not Reported | 2 | 1 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White/Caucasian | 147 | 51 | 44 | 242
  Race: Black or African American | 6 | 2 | 4 | 12
  Race: Asian | 2 | 0 | 0 | 2
  Race: American Indian or Alaska Native | 1 | 0 | 0 | 1
  Race: Hispanic | 1 | 0 | 0 | 1
  Race: Unknown | 8 | 3 | 5 | 16

OUTCOME MEASURES:

1. Primary Outcome: Phase 2: Complete Response (CR) Rate as Per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) 2018 Criteria
Description: CR rate=percent of participants who achieved CR or complete response with incomplete marrow recovery(CRi).CR=no evidence of new disease,absolute lymphocyte count(ALC) in peripheral blood<4x10^9 per liter(/L),regression of nodal masses to normal size <1.5 centimeters(cm) in longest diameter(LD),normal spleen and liver size,no constitutional symptoms,cytological/pathological evaluation of bone marrow(BM) smear/biopsy must be at least normocellular for age without evidence for typical chronic lymphocytic leukemia(CLL)/small lymphocytic lymphoma(SLL) lymphocytes by morphological criteria,peripheral blood counts with absolute neutrophil count(ANC)≥1.5x10^9/L or platelet≥100x10^9/L or hemoglobin≥110 grams per liter(g/L) without red blood cell(RBC) transfusions,all without need for exogenous growth factors.CRi=all CR criteria but with persistent anemia,thrombocytopenia,or neutropenia or hypocellular BM that is related to prior/ongoing drug toxicity(and not to CLL/SLL).
Time Frame: Up to 43.2 months
Population: ITT population for Phase 2 consisted of all participants who received at least one dose of each study drug (ublituximab, umbralisib, and venetoclax). Percentages were rounded off to the nearest decimal point.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V)
Number analyzed (Participants) | 149
percentage of participants | 33.6

2. Primary Outcome: Phase 2: Overall Response Rate (ORR) Per iwCLL 2018 Criteria
Description: ORR=percent of participants who achieve CR,CRi,partial response(PR) or PR with lymphocytosis(PR-L).CR=no evidence of new disease;ALC<4x10^9/L;regression of nodal masses to<1.5cm LD;normal spleen,liver size;no constitutional symptoms;cytological/pathological evaluation of BM smear/biopsy must be at least normocellular for age;ANC≥1.5x10^9/L,platelet≥100x10^9/L,Hb≥110g/L.CRi=CR criteria but with persistent anemia,thrombocytopenia,or neutropenia/hypocellular BM related to prior/ongoing drug toxicity.PR=no evidence of new disease,meets≥2 criteria:≥50% decrease from baseline(BL) in ALC(or decrease to<4x10^9/L) or sum of products(SPD) of target nodal lesions or CLL/SLL marrow infiltrate/Blymphoid;no target,splenic,liver,or non-target disease with worsening that meets criteria for definitive progressive disease(PD);platelet>100x10^9/L or Hb≥110g/L or ≥50% increase from BL in each.PR-L=PR criteria but not had ≥50% decrease from BL in ALC/decrease to<4x10^9/L.
Time Frame: Up to 43.2 months
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V)
Number analyzed (Participants) | 149
percentage of participants | 93.3

3. Primary Outcome: Phase 3: Progression-Free Survival (PFS) Per iwCLL 2018 Criteria
Description: PFS was assessed in participants treated with U2-V compared with U2. PFS was defined as the interval between randomization and the date of definitive PD (as confirmed by the IRC) or death due to any cause, whichever occurs first. Participants who had no event (progression or death) were censored at the day of their last adequate disease assessment. PD= appearance of new nodes >1.5 cm in the LD, >50% increase in greatest diameter, new or recurrent hepatomegaly or splenomegaly, new unequivocal extra-nodal lesion, new non-target disease, ≥50% increase from the nadir in the sum of products of diameters (SPD) of target lesions, ≥50% increase in the LD of an individual node or extra-nodal mass, splenic/hepatic enlargement of ≥50% from nadir, unequivocal increase in the size of non-target disease, transformation to a more aggressive histology, decrease in platelet count or Hgb, >50% decrease from the highest on-study platelet count, >20 g/L decrease from the highest on-study Hgb.
Time Frame: Up to 43.2 months
Population: ITT population for Phase 3 consisted of all participants who were randomized. Percentages were rounded off to the nearest decimal point.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
Number analyzed (Participants) | 56 | 56
months | NA [0.0 to 15.7] — Median was not estimable due to low number of participants with events. | NA [0.0 to 13.1] — Median was not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) vs Phase 3: Ublituximab + Umbralisib (U2); Test type: Superiority; p = 0.6960, Log Rank; Hazard Ratio (HR) = 0.778, 95% CI 2-sided [0.219 to 2.755]

4. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: The MRD negativity rate was defined as the percentage of participants who achieved MRD negative status post-baseline, defined as a quantitative detection of less than one CLL/SLL cell in 10000 leukocytes by flow cytometry (MRD level, 10^-4) in blood or bone marrow (BM). If a participant was determined to be MRD negative by peripheral blood, a bone marrow aspirate was obtained to assess MRD in the bone marrow. Participants who did not have an MRD assessment at any post-baseline visits were considered non-responders and were included in the denominator when calculating MRD negativity rate.
Time Frame: Up to 43.2 months
Population: In Phase 2, ITT population consisted of all participants who received at least one dose of each study drug (ublituximab, umbralisib, and venetoclax); and in Phase 3, ITT population consisted of all participants who were randomized. Percentages were rounded off to the nearest decimal point.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
Number analyzed (Participants) | 149 | 56 | 56
percentage of participants | 94.0 [88.8 to 97.2] | 50.0 [36.3 to 63.7] | 19.6 [10.2 to 32.4]

5. Secondary Outcome: Number of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product. An AE does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is any AE that occur after first dosing of study medication and through the end of the study or through 30 days after the last dose of study treatment, or is considered treatment-related regardless of the start date of the event, or is present before first dosing of study medication but worsens in intensity or the investigator subsequently considers treatment-related.
Time Frame: Up to 43.2 months
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
Number analyzed (Participants) | 165 | 56 | 53
Participants | 165 | 56 | 51

6. Secondary Outcome: Phase 2: Time to Response (TTR) Per iwCLL 2018 Criteria
Description: TTR was defined as the interval from enrollment to first documentation of CR, CRi, PR, or PR-L. TTR was analyzed via Kaplan-Meier method. CR=no evidence of new disease; ALC<4x10^9/L; regression of nodal masses to <1.5cm LD; normal spleen ,liver size; no constitutional symptoms; cytological/pathological evaluation of BM smear/biopsy must be at least normocellular for age; ANC≥1.5x10^9/L, platelet≥100x10^9/L, Hb≥110g/L. CRi=CR criteria but with persistent anemia, thrombocytopenia, or neutropenia/hypocellular BM related to prior/ongoing drug toxicity.PR=no evidence of new disease,meets≥2 criteria:≥50% decrease from BL in ALC (or decrease to<4x10^9/L) or SPD of target nodal lesions or CLL/SLL marrow infiltrate/B-lymphoid; no target, splenic, liver, or non-target disease with worsening that meets criteria for definitive PD; platelet>100x10^9/L or Hb≥110g/L or ≥50% increase from BL in each.PR-L=PR criteria but not had ≥50% decrease from BL in ALC/decrease to<4x10^9/L.
Time Frame: Up to 43.2 months
Population: ITT population for Phase 2 consisted of all participants who received at least one dose of each study drug (ublituximab, umbralisib, and venetoclax). Only responders i.e., participants with ORR were assessed for this outcome measure.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V)
Number analyzed (Participants) | 139
months | 2.6 [2.3 to 18.5]

7. Secondary Outcome: Phase 2: Duration of Response (DOR) Per iwCLL 2018 Criteria
Description: DOR=interval from 1st documentation of CR,CRi,PR or PR-L to earlier of 1st documentation of definitive PD or death from any cause.CR=no evidence of new disease;ALC<4x10^9/L;regression of nodal masses to<1.5cm LD;normal spleen,liver size;no constitutional symptoms;cytological/pathological evaluation of BM smear/biopsy must be at least normocellular for age;ANC≥1.5x10^9/L,platelet≥100x10^9/L,Hb≥110g/L.CRi=CR criteria but with persistent anemia,thrombocytopenia,neutropenia/hypocellular BM related to prior/ongoing drug toxicity.PR=no evidence of new disease,meets≥2 criteria:≥50% decrease from BL in ALC(or decrease to<4x10^9/L) or SPD of target nodal lesions or CLL/SLL marrow infiltrate/Blymphoid;no target,splenic,liver,or non-target disease with worsening that meets criteria for definitive PD;platelet>100x10^9/L or Hb≥110g/L or ≥50% increase from BL in each.PR-L=PR criteria;not≥50% decrease from BL in ALC/decrease to<4x10^9/L.PD=evidence of new disease per protocol-specififed criteria.
Time Frame: Up to 43.2 months
Population: as for outcome 6
Measure: Median (Full Range); unit: months
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V)
Number analyzed (Participants) | 139
months | 21.1 [0.0 to 24.8]

8. Secondary Outcome: Phase 3: CR Rate as Assessed by an Independent Review Committee (IRC) Per iwCLL 2018 Criteria
Description: CR rate=percent of participants who achieved CR or CRi. CR=no evidence of new disease; ALC<4x10^9/L; regression of nodal masses to <1.5 cm LD; normal spleen, liver size; no constitutional symptoms; cytological/pathological evaluation of BM smear/biopsy must be at least normocellular for age; ANC ≥1.5x10^9/L, platelet ≥100x10^9/L, Hb ≥110g/L. CRi=CR criteria but with persistent anemia,thrombocytopenia,or neutropenia/hypocellular BM related to prior/ongoing drug toxicity. CR assessment was subject to independent confirmation by the IRC in participants enrolled to the Phase 3 stage of the study.
Time Frame: Up to 43.2 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
Number analyzed (Participants) | 56 | 56
percentage of participants | 17.9 | 8.9

9. Secondary Outcome: Phase 3: ORR as Assessed by IRC Per iwCLL 2018 Criteria
Description: ORR=percent of participants who achieve CR, CRi, PR or PR-L.CR=no evidence of new disease; ALC<4x10^9/L; regression of nodal masses to<1.5cm LD; normal spleen and liver size; no constitutional symptoms; cytological/pathological evaluation of BM smear/biopsy must be at least normocellular for age; ANC≥1.5x10^9/L, platelet≥100x10^9/L, Hb≥110g/L. CRi=CR criteria but with persistent anemia, thrombocytopenia, or neutropenia/hypocellular BM related to prior/ongoing drug toxicity.PR=no evidence of new disease,meets≥2 criteria:≥50% decrease from baseline (BL) in ALC (or decrease to<4x10^9/L) or SPD of target nodal lesions or CLL/SLL marrow infiltrate/B-lymphoid; no target, splenic, liver, or non-target disease with worsening that meets criteria for definitive PD; platelet>100x10^9/L or Hb≥110g/L or ≥50% increase from BL in each.PR-L=PR criteria but not had ≥50% decrease from BL in ALC/decrease to<4x10^9/L.
Time Frame: Up to 43.2 months
Population: as for outcome 3
Measure: Number; unit: percentage of participants
Arm/Group | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
Number analyzed (Participants) | 56 | 56
percentage of participants | 71.4 | 62.5

10. Secondary Outcome: Phase 3: Overall Survival (OS)
Description: Overall Survival (OS) was defined as the interval from randomization to death from any cause. OS data was censored at the last documented date that the participant was confirmed alive for participants who withdrew consent or were lost to follow-up prior to the end of the study, and for participants whose vital status in the study could not be determined.
Time Frame: Up to 43.2 months
Population: ITT population for Phase 3 consisted of all participants who were randomized.
Measure: Median (Full Range); unit: months
Arm/Group | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
Number analyzed (Participants) | 56 | 56
months | NA [0.5 to 16.6] — Median was not estimable due to low number of participants with event. | NA [0.0 to 16.2] — Median was not estimable due to low number of participants with event.
Statistical Analysis 1: Comparison: Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) vs Phase 3: Ublituximab + Umbralisib (U2); Test type: Superiority; p = 0.1038, Log Rank; Hazard Ratio (HR) = 0.201, 95% CI 2-sided [0.023 to 1.721]

ADVERSE EVENTS:
Time Frame: Up to 43.2 months
Description: All-Cause Mortality for Phase 3: ITT population consisted of all participants who were randomized; All-Cause Mortality (Phase 2 arm); Serious and Other Adverse Events: Safety population consisted of all participants who received at least one dose of any study drug (ublituximab, umbralisib, and venetoclax).
Arm/Group | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) | Phase 3: Ublituximab + Umbralisib (U2)
All-Cause Mortality (participants affected / at risk) | 32/165 | 1/56 | 5/56
Serious Adverse Events (participants affected / at risk) | 84/165 | 12/56 | 16/53
Other Adverse Events (participants affected / at risk) | 165/165 | 56/56 | 49/53
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) (N=165) | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) (N=56) | Phase 3: Ublituximab + Umbralisib (U2) (N=53)
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 2 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 5 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Pericarditis (Cardiac disorders) | 1 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 7 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 3 | 1 | 1
Death (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 0
Acute on chronic liver failure (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 1
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1 | 0
Liver injury (Hepatobiliary disorders) | 0 | 0 | 1
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 0 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 0 | 1
COVID-19 (Infections and infestations) | 15 | 0 | 3
COVID-19 pneumonia (Infections and infestations) | 13 | 2 | 4
Pneumonia (Infections and infestations) | 9 | 2 | 2
Sepsis (Infections and infestations) | 3 | 0 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 2 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Candida infection (Infections and infestations) | 1 | 0 | 0
Hepatitis B reactivation (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 1 | 0 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia legionella (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Pneumonia viral (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 2 | 1 | 2
Accidental overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Platelet count decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 0 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
T-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Intestinal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Dural arteriovenous fistula (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 5 | 0 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Reproductive system and breast disorders) | 0 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 2: Ublituximab + Umbralisib + Venetoclax (U2-V) (N=165) | Phase 3: Ublituximab + Umbralisib + Venetoclax (U2-V) (N=56) | Phase 3: Ublituximab + Umbralisib (U2) (N=53)
Anaemia (Blood and lymphatic system disorders) | 36 | 5 | 4
Neutropenia (Blood and lymphatic system disorders) | 31 | 11 | 5
Lymphadenopathy (Blood and lymphatic system disorders) | 11 | 1 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 3 | 3
Leukocytosis (Blood and lymphatic system disorders) | 3 | 3 | 0
Palpitations (Cardiac disorders) | 12 | 2 | 0
Tinnitus (Ear and labyrinth disorders) | 11 | 2 | 2
Vision blurred (Eye disorders) | 12 | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 120 | 30 | 23
Nausea (Gastrointestinal disorders) | 94 | 26 | 27
Abdominal pain (Gastrointestinal disorders) | 32 | 3 | 5
Vomiting (Gastrointestinal disorders) | 27 | 6 | 6
Constipation (Gastrointestinal disorders) | 26 | 7 | 7
Dyspepsia (Gastrointestinal disorders) | 20 | 3 | 5
Abdominal distension (Gastrointestinal disorders) | 16 | 3 | 2
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 14 | 3 | 5
Stomatitis (Gastrointestinal disorders) | 12 | 3 | 1
Flatulence (Gastrointestinal disorders) | 10 | 0 | 2
Abdominal pain upper (Gastrointestinal disorders) | 8 | 1 | 3
Dry mouth (Gastrointestinal disorders) | 6 | 3 | 0
Toothache (Gastrointestinal disorders) | 3 | 3 | 0
Fatigue (General disorders) | 74 | 25 | 17
Oedema peripheral (General disorders) | 32 | 6 | 6
Pyrexia (General disorders) | 28 | 8 | 4
Chills (General disorders) | 21 | 3 | 2
Generalised oedema (General disorders) | 0 | 3 | 1
COVID-19 (Infections and infestations) | 31 | 6 | 2
Upper respiratory tract infection (Infections and infestations) | 14 | 0 | 2
Pneumonia (Infections and infestations) | 13 | 2 | 2
Urinary tract infection (Infections and infestations) | 13 | 2 | 0
Sinusitis (Infections and infestations) | 8 | 3 | 4
Candida infection (Infections and infestations) | 5 | 3 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 112 | 38 | 26
Contusion (Injury, poisoning and procedural complications) | 17 | 2 | 2
Neutrophil count decreased (Investigations) | 77 | 20 | 10
Platelet count decreased (Investigations) | 34 | 6 | 4
Aspartate aminotransferase increased (Investigations) | 33 | 12 | 15
Alanine aminotransferase increased (Investigations) | 31 | 10 | 17
White blood cell count decreased (Investigations) | 27 | 4 | 1
Blood creatinine increased (Investigations) | 13 | 7 | 4
Blood alkaline phosphatase increased (Investigations) | 10 | 1 | 3
Lymphocyte count decreased (Investigations) | 9 | 1 | 1
Blood bilirubin increased (Investigations) | 8 | 2 | 5
Blood lactate dehydrogenase increased (Investigations) | 8 | 6 | 1
Weight decreased (Investigations) | 8 | 2 | 4
Decreased appetite (Metabolism and nutrition disorders) | 41 | 4 | 6
Hypokalaemia (Metabolism and nutrition disorders) | 24 | 3 | 3
Dehydration (Metabolism and nutrition disorders) | 16 | 2 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 14 | 3 | 2
Hypocalcaemia (Metabolism and nutrition disorders) | 13 | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 11 | 1 | 2
Hyperuricaemia (Metabolism and nutrition disorders) | 11 | 3 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 2 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 3 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 41 | 5 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 8 | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 0 | 3
Muscle spasms (Musculoskeletal and connective tissue disorders) | 14 | 4 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 14 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 11 | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 9 | 3 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 5 | 3 | 1
Dizziness (Nervous system disorders) | 43 | 9 | 9
Headache (Nervous system disorders) | 43 | 15 | 13
Dysgeusia (Nervous system disorders) | 19 | 7 | 2
Tremor (Nervous system disorders) | 13 | 2 | 1
Paraesthesia (Nervous system disorders) | 9 | 0 | 2
Insomnia (Psychiatric disorders) | 47 | 16 | 12
Anxiety (Psychiatric disorders) | 14 | 7 | 3
Depression (Psychiatric disorders) | 7 | 3 | 2
Pollakiuria (Renal and urinary disorders) | 13 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 38 | 9 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 33 | 8 | 8
Productive cough (Respiratory, thoracic and mediastinal disorders) | 10 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 9 | 3 | 5
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 7 | 4 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 4
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 16 | 5 | 6
Rash (Skin and subcutaneous tissue disorders) | 14 | 7 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 13 | 0 | 3
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 5 | 4
Alopecia (Skin and subcutaneous tissue disorders) | 10 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 9 | 2 | 4
Night sweats (Skin and subcutaneous tissue disorders) | 6 | 3 | 3
Hypertension (Vascular disorders) | 20 | 3 | 2
Hypotension (Vascular disorders) | 11 | 1 | 2
Flushing (Vascular disorders) | 10 | 1 | 3

LIMITATIONS AND CAVEATS:
Due to sponsor's business decision, the clinical trial was terminated by the sponsor prematurely. As such, the study results are reflective of the data captured to the time of study termination and with limited data verification.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-05): https://cdn.clinicaltrials.gov/large-docs/25/NCT03801525/Prot_SAP_000.pdf